CLINICAL TRIAL: NCT03197025
Title: A Phase I Study of Immunotherapy With E6 T Cell Receptor T Cells for Vulvar High-Grade Squamous Intraepithelial Lesions
Brief Title: Immunotherapy With E6 T Cell Receptor (TCR) T Cells for Vulvar High-Grade Squamous Intraepithelial Lesions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was closed due to investigator discretion based on the lack of perceived clinical activity observed in the study.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott Norberg, D.O., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170116; 17-C-0116
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Human Papillomavirus; HPV-16; High Grade Squamous Intraepithelial Lesion
Keywords: HPV-16; Premalignancy; T Cell Therapy
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Arm 1 - Dose Escalation (Experimental): Patients will undergo leukapheresis, then treatment with E6 T Cell Receptor (TCR) cells (at escalating doses) + aldesleukin
  Interventions: Drug: Aldesleukin; Biological: E6 T Cell Receptor (TCR)
- 2/Arm 2 - Maximum Tolerated Dose (MTD) (Experimental): Patients will undergo leukapheresis, then treatment with E6 T Cell Receptor (TCR) cells (at the MTD) + aldesleukin
  Interventions: Drug: Aldesleukin; Biological: E6 T Cell Receptor (TCR)

INTERVENTIONS:
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg (based on total body weight) intravenous (IV) infused over 15 minutes approximately every 12 hours for a maximum of two doses.
  Other Names: Interleukin-2
Biological: E6 T Cell Receptor (TCR) — On day 0, the E6 TCR cells will be administered one time, intravenously over 20 to 30 minutes

SUMMARY:
Background:

Vulvar high-grade squamous intraepithelial lesion (HSIL) is caused by infection of the vulva with human papillomavirus (HPV). In a small percentage of cases, vulvar HSIL can turn into cancer. The risk of cancer can be reduced by treating HSIL. A personalized immune treatment might rid the body of HPV infection and thereby cure vulvar HSIL. The immune treatment in this study is called T cell therapy. The cells are E6 T Cell Receptor (TCR) T cells. Participants will also get aldesleukin (IL-2) to help the cells last longer.

Objective:

To find a safe dose of E6 TCR T cells combined with aldesleukin to use in people with vulvar HSIL.

Eligibility:

Design:

Participants will be screened with:

Physical exam

Medical history

Blood, lab, and pregnancy tests

Heart tests

Chest x-ray

Sample of tissue taken from the vulva (biopsy).

Participants will have leukapheresis. Blood will be removed by a needle in one arm. A machine removes white blood cells from the blood. The rest of the blood is returned by needle in the other arm. The white blood cells will be changed into E6 TCR T cells and grown in a lab. About 3 weeks later, participants will be admitted to the hospital for about 5 days. They will get the cells through a tube placed in a vein. They will get IL-2 the same way. Participants will recover 1-3 days in the hospital. They will be monitored closely. They will have blood and lab tests. Participants will have follow-up visits with lab tests and a physical exam every few months for 5 years. At some visits they will also have leukapheresis, blood tests, or vulvar biopsy.

DETAILED DESCRIPTION:
Background:

* Vulvar high-grade squamous intraepithelial lesion (HSIL) is a premalignant epithelial lesion that is frequently multifocal and/or recurrent.
* The primary treatment is surgery, which may result in disfigurement and compromise of the urethra, anus, or clitoris. Recurrence after surgery is common and primarily treated with additional surgery.
* Vulvar HSIL is caused by chronic infection with the human papillomavirus (HPV) type 16 infection. In this clinical trial the HPV-16 infection is targeted with a single infusion of autologous T cells that have been genetically engineered to express an HPV-16 E6-specific

T cell receptor (E6 TCR T cells).

Objective:

-Determine the safety of E6 TCR T cells for the treatment of vulvar HSIL.

Eligibility:

* Histologically confirmed diagnosis of HPV-16+ vulvar HSIL.
* Expression of the human leukocyte antigen (HLA)-A2*02:01 allele.
* Measurable lesion(s) that are recurrent or cannot be resected with acceptable cosmetic or functional results.
* Age greater than or equal to 18 years old and less than or equal to 65 years old.
* Eastern Oncology Cooperative Group Performance Score of 0 or 1.

Design:

* This is a phase I clinical trial with a 3+3 dose escalation design.
* Subjects will receive E6 TCR T cells followed by up to two doses of aldesleukin 720,000 IU/kg intravenous (IV).
* No conditioning regimen will be given, aldesleukin will be capped at a maximum of two doses, and E6 TCR T cell dosing will begin at dose level -1 from the previously determined safe dose.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have vulvar High-Grade Squamous Intraepithelial Lesions (HSIL) as confirmed by pathology report from a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
  2. Vulvar HSIL must be human papilloma virus (HPV)-16+ by a polymerase chain reaction (PCR), ribonucleic acid (RNA), or in situ hybridization test from a CLIA certified laboratory.
  3. Patients must have measurable lesion(s) as defined in section 6.3.2 and one or more of the following criteria:

     1. Failure of surgery to control disease (i.e. positive margins or recurrence of HSIL after surgery).
     2. Multifocal or extensive disease for which surgery would result in major deformity that is not be acceptable to the patient.
     3. Disease for which surgery would have a risk of functional impairment that is not be acceptable to the patient (i.e. involve partial or complete excision of the clitoris, anus, vagina, or urethra).
  4. Patients may have received any previous therapy, including surgical excision, but must have histologically documented recurrence on new biopsy and a measurable lesion that meets the above criteria.
  5. The presence of disease that can be biopsied for research purposes is not an inclusion criterion.
  6. Patients must have the human leukocyte antigen (HLA)-A*02:01 allele
  7. Age greater than or equal to 18 years and less than or equal to 65 years. As age increases, the ability to tolerate the toxicities of aldesleukin decreases, so the patient population for this study will include up to and including 60 years of age to increase safety.
  8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. Able to understand and sign the Informed Consent Document.
  9. Women of child-bearing potential must have a negative pregnancy test. Women of child-bearing potential are defined as all women who are not post-menopausal or who have not had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
  10. The effects of E6 T Cell Receptor (TCR) T Cells on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
  11. Seronegative for human immunodeficiency virus (HIV) antibody. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment.
  12. Seronegative for hepatitis B antigen and hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by reverse transcription (RT)-PCR and be hepatitis C virus (HCV) RNA negative.
  13. Must be willing to participate in Gene Therapy Long Term Followup Protocol (15-C-0141), which will follow patients for up to 15 years per Food and Drug Administration (FDA) requirements.
  14. Patients must have normal organ and marrow function as defined below:
* leukocytes greater than or equal to 3,000/mcL
* absolute neutrophil count greater than or equal to 1,000/mcL
* platelets greater than or equal to 150,000/mcL
* hemoglobin greater than or equal to 10.0 g/dL
* total bilirubin within normal institutional limits except in patients with Gilbert's Syndrome who must have a total bilirubin < 3.0 mg/dL
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) Serum ALT/AST < 3 times ULN
* creatinine less than 1.5 times baseline, < 1.5 times upper limit of normal (ULN)

OR

-creatinine clearance less than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal (by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)

EXCLUSION CRITERIA:

1. Patients who are receiving any other investigational agents
2. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E6 TCR, breastfeeding should be discontinued if the mother is treated with E6 TCR. These potential risks may also apply to other agents used in this study.
3. Uncontrolled intercurrent illness including, but not limited to, any ongoing or active infection (e.g. requiring anti-infective therapy), coagulation disorders, cardiovascular disorders, respiratory disorders, cancer, or psychiatric illness/social situations (within the last six months) that would limit compliance with study requirements.
4. Any form of systemic immunodeficiency, including acquired deficiency such as HIV or primary immunodeficiency such as Severe Combined Immunodeficiency Disease. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the treatment.
5. Concurrent systemic steroid therapy if greater than the equivalent of 5 mg prednisone by mouth (PO) daily. Patients previously on steroids must be off steroids for four weeks prior to treatment.
6. Any history of clinically significant cardiac arrhythmia, coronary revascularization, ischemic symptoms, or previously documented left ventricular ejection fraction (LVEF) of less than or equal to 45%. A cardiac stress test is required for all patients greater than 50 years old. A cardiac stress test may also be performed for any clinical concern. Patients with cardiac ischemia are not eligible.
7. Patients with any active invasive cancer are not eligible.
8. Patients vulvar HSIL that is not HPV-16+ or is associated with multiple types of high-risk HPV are not eligible.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Norberg, DO, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0116.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one participant was enrolled, thus Arm/Group - 2/Arm 2 MTD was not done.
Groups:
- Dose Level -1: 0.7 x 10^10 Transduced T Cells: Patients will undergo leukapheresis, then treatment with E6 T Cell Receptor (TCR) cells (at escalating doses) + aldesleukin
  Aldesleukin: Aldesleukin 720,000 IU/kg (based on total body weight) intravenous (IV) infused over 15 minutes approximately every 12 hours for a maximum of two doses.
  E6 T Cell Receptor (TCR): On day 0, the E6 TCR cells will be administered one time, intravenously over 20 to 30 minutes
Period: Overall Study
Arm/Group | Dose Level -1: 0.7 x 10^10 Transduced T Cells
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One participant was enrolled, thus Arm/Group - 2/Arm 2 MTD was not done.
Arm/Group | Dose Level -1: 0.7 x 10^10 Transduced T Cells
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of E6 T Cell Receptor (TCR) T Cells for the Treatment of Vulvar High-Grade Squamous Intraepithelial Lesions (HSIL)
Description: MTD is defined as the highest dose at which a maximum of 1 of 6 participants has a dose limiting toxicity (DLT). A DLT is defined as all treatment related Grade 3 (i.e. severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living (ADL)) and greater adverse events occurring within 30 days of the cell infusion with the exception of Grade 3 fever or chills responsive to symptomatic treatment that resolve to ≤ grade 2 in 48 hours. Grade 3 hypotension or oliguria responsive to ≤ 1.5L of intravenous fluid boluses in 24 hours that resolves to ≤ grade 2 in 48 hours. Grade 3 dyspnea/hypoxia that improves to ≤ grade 2 or less with supplemental oxygen and resolves to ≤ grade 2 without supplemental oxygen in 48 hours. Grade 3 creatinine or electrolyte abnormalities that resolve to ≤ grade 2 in 48 hours.
Time Frame: within 30 days of cell infusion
Measure: Number; unit: cells
Arm/Group | Dose Level -1: 0.7 x 10^10 Transduced T Cells
Number analyzed (Participants) | 1
cells | NA — One patient was analyzed in an attempt to determine the MTD. However, since there was only one patient treated, the primary outcome cannot be measured (since the outcome was determining the MTD).

2. Secondary Outcome: Number of Participants With a Clinical Response Treated With E6 T Cell Receptor (TCR) T Cells for Vulvar High-Grade Squamous Intraepithelial Lesions (HSIL)
Description: Complete Response (CR) is disappearance of all target lesions. No appearance of new lesions. Partial Response (PR) is a ≥50% decrease in the sum of the product of the longest perpendicular diameters of target lesions, taking as reference the baseline measurements. No appearance of new lesions. No increase of greater than 25% of index lesion. Progressive disease is a ≥25% increase in the sum of the product of the longest perpendicular diameters of target lesions, taking as reference the smallest product on study (this includes the baseline product if that is the smallest on study). In addition to the relative increase of 25%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progression. Non-CR/Non-PD is neither sufficient decrease to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest product of diameters while on study.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level -1: 0.7 x 10^10 Transduced T Cells
Number analyzed (Participants) | 1
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Progressive Disease (PD) | 0
  Non-CR/Non-PD | 1

3. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 4 months and 17 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level -1: 0.7 x 10^10 Transduced T Cells
Number analyzed (Participants) | 1
Participants | 1

4. Other Pre Specified Outcome: Number of Grade 4 Lymphocyte Count Decreased Dose Limiting Toxicities (DLT)
Description: DLT is defined as all treatment related Grade 3 (severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living (ADL) and greater adverse events occurring within 30 days of the cell infusion with the exception of the following expected transient effects of aldesleukin. Grade 3 fever or chills responsive to symptomatic treatment that resolve to ≤ grade 2 in 48 hours. Grade 3 hypotension or oliguria responsive to ≤ 1.5L of intravenous fluid boluses in 24 hours that resolves to ≤ grade 2 in 48 hours. Grade 3 dyspnea/hypoxia that improves to ≤ grade 2 or less with supplemental oxygen and resolves to ≤ grade 2 without supplemental oxygen in 48 hours. Grade 3 creatinine or electrolyte abnormalities that resolve to ≤ grade 2 in 48 hours.
Time Frame: within 30 days of cell infusion
Population: The protocol was amended to exclude Grade 3 or higher white blood cell count decreased/lymphocyte count decreased that resolved to less than Grade 2 in 72 hours. This was done since transient lymphopenia is not a clinically significant event.
Measure: Number; unit: Toxicities
Arm/Group | Dose Level -1: 0.7 x 10^10 Transduced T Cells
Number analyzed (Participants) | 1
Toxicities | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 4 months and 17 days.
Description: One participant was enrolled, thus Arm/Group - 2/Arm 2 MTD was not done.
Arm/Group | Dose Level -1: 0.7 x 10^10 Transduced T Cells
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level -1: 0.7 x 10^10 Transduced T Cells (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT03197025/Prot_SAP_000.pdf
  • Informed Consent Form: Standard consent (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03197025/ICF_001.pdf
  • Informed Consent Form: Screening consent (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03197025/ICF_002.pdf